CLINICAL TRIAL: NCT02235246
Title: The Effect of Perioperative Intravenous Magnesium on Pain After Endoscopic Submucosal Dissection for Gastric Neoplasm: Prospective Randomized Double-blind Placebo Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2014-0601
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Neoplasm
Keywords: perioperative intravenous magnesium; endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Experimental)
  Interventions: Drug: Normal saline
- magnesium sulfate (Active Comparator)
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — magnesium sulfate 50 mg/kg will be administrated during 10 min before anesthetic induction in patients undergoing endoscopic submucosal dissection.
  Arms: magnesium sulfate
Drug: Normal saline — Normal saline will be administrated during 10 min before anesethetic induction in patients undergoing endoscopic submucosal dissection.
  Arms: normal saline

SUMMARY:
Endoscopic submucosal dissection (ESD) is an effective treatment for early gastric cancer or premalignant lesions in the stomach. ESD enables en bloc resection of gastrointestinal neoplasms, increases the rates of histologically complete resections, and also reduces local recurrence rates. Despite these advantages, ESD is thought to induce various complications. Wellknown ESD-related complications include perforation, postoperative bleeding, or stricture. In addition, minor adverse events after ESD are also commonly noticed. Pain is one of these frequently noticed minor ESD related complications, is the main reason for prolongation of the hospital stay, and is related to patients' compliance; however, there is a tendency to neglect or underestimate post-ESD pain. The causes of pain associated with ESD are thought to be associated with transmural burn or transmural air leak. Some studies have tried to control localized pain during and after ESD using local lidocaine, single dose postoperative intravenous dexamethasone or a transdermal fentanyl patch. Magnesium has been reported to alter the perception and duration of pain and produce important analgesic effects. It is included the suppression of neuropathic pain, potentiation of morphine analgesia, and attenuation of morphine tolerance. Although the exact mechanism is not yet fully understood, the analgesic properties of magnesium are believed to stem from regulation of calcium influx into the cell and antagonism of N-methyl-D-aspartate receptors in the central nervous system. Also, magnesium may prolong neuromuscular blockade after administration of neuromuscular blocking drugs, increase sedation and contribute to serious cardiac morbidity. And magnesium as a hypotensive anaesthesia technique supply objectively better operative field, reduction in the duration of surgery and reduced blood loss. There have been no previous trials on the use of magnesium specifically for pain control following ESD. Thus, the purpose of this study was to assess the efficacy of intravenous magnesium for pain relief after ESD.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1~2, 2. age of 40- 80 years

Exclusion Criteria:

1. patients who cannot read,
2. patients refusing the study
3. allergy to magnesium
4. chronic pain
5. chronic abuse of opioid or NSAID
6. neuromuscular block
7. atrioventricular conductance block
8. liver failure,

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
pain score | average 24hours from endoscopic processure
  Pain score related with endoscopic mucosal resection will be evaluated with numerical rating scale (0 ~ 10) at time of 30 min, 1 hr, 6 hr, and 24 hr after procedure end.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JE, Shin CS, Lee YC, Lee HS, Ban M, Kim SY. Beneficial effect of intravenous magnesium during endoscopic submucosal dissection for gastric neoplasm. Surg Endosc. 2015 Dec;29(12):3795-802. doi: 10.1007/s00464-015-4514-1. Epub 2015 Sep 3. PMID 26335078